CLINICAL TRIAL: NCT04625270
Title: A Phase 2 Study of Avutometinib (VS-6766) (Dual RAF/MEK Inhibitor) Alone and In Combination With Defactinib (FAK Inhibitor) in Recurrent Low-Grade Serous Ovarian Cancer (LGSOC)
Brief Title: A Study of Avutometinib (VS-6766) v. Avutometinib (VS-6766) + Defactinib in Recurrent Low-Grade Serous Ovarian Cancer With and Without a KRAS Mutation
Acronym: RAMP 201
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VS-6766-201; GOG-3052 (Other: The GOG Foundation, Inc.); ENGOT-ov60 (Other: ENGOT)
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-03

CONDITIONS: Low Grade Ovarian Serous Adenocarcinoma; Ovarian Cancer
Keywords: Low Grade Serous Ovarian Cancer; KRAS, KRAS wt
MeSH Terms: conditions — Ovarian Neoplasms | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A (Experimental): To determine the optimal regimen, either avutometinib(VS-6766) monotherapy or avutometinib (VS-6766) in combination with defactinib, for subsequent evaluation for efficacy in the Expansion Phase (Part B)
  Interventions: Drug: avutometinib (VS-6766); Drug: avutometinib (VS-6766) and defactinib
- Part B (Experimental): To determine the efficacy of the optimal regimen identified from Part A
  Interventions: Drug: avutometinib (VS-6766); Drug: avutometinib (VS-6766) and defactinib
- Part C: (Experimental): To evaluate additional efficacy parameters for the optimal regimen identified in Part A.
  Interventions: Drug: avutometinib (VS-6766) and defactinib
- Part D (Experimental): To evaluate additional efficacy parameters for a lower dose of avutometinib in combination with defactinib
  Interventions: Drug: avutometinib (VS-6766) and defactinib

INTERVENTIONS:
Drug: avutometinib (VS-6766) — avutometinib (VS-6766) monotherapy
  Arms: Part A; Part B
Drug: avutometinib (VS-6766) and defactinib — avutometinib (VS-6766) and defactinib combination
  Other Names: avutometinib (VS-6766) and VS-6063

SUMMARY:
This study will assess the safety and efficacy of avutometinib (VS-6766) monotherapy and in combination with defactinib in subjects with recurrent Low-Grade Serous Ovarian Cancer (LGSOC)

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label Phase 2 study designed to evaluate safety and tolerability and preliminary efficacy of avutometinib (VS-6766) versus avutometinib (VS-6766) in combination with defactinib in subjects with molecularly profiled recurrent LGSOC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven LGSOC (ovarian, peritoneal)
* Progression or recurrence of LGSOC after at least one prior systemic therapy for metastatic disease.
* Measurable disease according to RECIST 1.1
* An Eastern Cooperative Group (ECOG) performance status ≤ 1.
* Adequate organ function
* Adequate recovery from toxicities related to prior treatments
* Agreement to use highly effective method of contraceptive, if necessary

Exclusion Criteria:

* Systemic anti-cancer therapy within 4 weeks of the first dose of study therapy
* Co-existing high-grade ovarian cancer or another histology
* History of prior malignancy with recurrence <3 years from the time of enrollment
* Major surgery within 4 weeks
* Symptomatic brain metastases requiring steroids or other interventions
* Known SARS-Cov2 infection (clinical symptoms) ≤28 days prior to first dose of study therapy
* For subjects with prior MEK exposure, Grade 4 toxicity deemed related to the MEK inhibitor
* Active skin disorder that has required systemic therapy within the past year
* History of rhabdomyolysis
* Concurrent ocular disorders
* Concurrent heart disease or severe obstructive pulmonary disease
* Subjects with the inability to swallow oral medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part A: Determine optimal regimen of avutometinib (VS-6766) monotherapy or in combination with defactinib | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1
Part B: To determine the efficacy of the optimal regimen identified from Part A | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1
Part C: To evaluate additional efficacy parameters for the optimal regimen identified in Part A | From start of treatment to confirmation of response; 24 weeks
  Confirmed overall response rate per RECIST 1.1
Part D:To evaluate additional efficacy parameters for a lower dose of avutometinib in combination with defactinib | From start of treatment to confirmation of response; 24 weeks
  Confirmed ORR defined according to RECIST 1.1

SECONDARY OUTCOMES:
Overall Response Rate as assessed by Investigator | From start of treatment to confirmation of response; 24 weeks
  Proportioned subjects achieving a CR or PR as assess by the investigator
Duration of Response (DOR) | Time from the first documentation of response to first documentation of progressive disease or death due to any cause, greater than or equal to 6 months
  From time of first response to PD as assessed by the BIRC
Disease Control Rate (DCR) | Greater than or equal to 8 weeks
  CR+PR+stable disease
Progression Free Survival (PFS) | Up to 5 years
  From time of first dose of study intervention to PD or death for any cause
Overall Survival (OS) | Up to 5 years
  From time of first dose of study intervention to death

CONTACTS AND LOCATIONS:
Overall Officials: Susana Banerjee, MBBS,MA,PhD, Principal Investigator — European Network of Gynaecological Oncological Trial Groups (ENGOT); Rachel Grisham, MD, Principal Investigator — GOG Foundation; MD Verastem, Study Director — Verastem, Inc.
Locations (47):
- United States (27):
  - Arizona Oncology Associates PC HAL, Scottsdale, Arizona
  - Sansum Clinic, Santa Barbara, California
  - Yale School of Medicine, New Haven, Connecticut
  - Advent Health, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute - Center for Women's Oncology, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Maryland Oncology and Hematology, P.A., Glenn Dale, Maryland
  - Minnesota Oncology Hematology PA, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Women's Health Institute, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology Austin Central, Austin, Texas
  - Texas Oncology- Dallas Presbyterian Hospital, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, Longview, Texas
  - Texas Oncology, McAllen, Texas
  - Texas Oncology, San Antonio, Texas
  - Texas Oncology, The Woodlands, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
- Belgium (3):
  - UZ Gent Medische Oncologie, Ghent
  - UZ Leuven, Leuven
  - CHU de Liege, Liège
- Canada (2):
  - Centre de recherche di Centre Hospitalier de i'Universite de Montreal, Montreal
  - Princess Margaret Cancer Centre, Toronto
- France (4):
  - Hopital Jean Minjoz, Besançon
  - Centre Leon Berard, Lyon
  - ICM - Val d'Aurelle, Montpellier
  - Institut Curie, Paris
- Italy (2):
  - Insituto Europeo di Oncologia I.R.C.C.S, Milan
  - U.O.C. Oncologia 2, Istituto Oncologico Veneto I.R.C.C.S., Padua
- Spain (4):
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (5):
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - UCLH Cancer Clinical Trials Unit, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee SN, Van Nieuwenhuysen E, Aghajanian C, D'Hondt V, Monk BJ, Clamp A, Prendergast E, Oaknin A, Ring K, Colombo N, Holloway RW, Rodrigues M, Chon HS, Gourley C, Santin AD, Thaker PH, Gennigens C, Newman G, Salinas E, Youssoufian H, Moore KN, Lustgarten S, O'Malley DM, Van Gorp T, Grisham RN. Efficacy and Safety of Avutometinib +/- Defactinib in Recurrent Low-Grade Serous Ovarian Cancer: Primary Analysis of ENGOT-OV60/GOG-3052/RAMP 201. J Clin Oncol. 2025 Sep;43(25):2782-2792. doi: 10.1200/JCO-25-00112. Epub 2025 Jul 11. PMID 40644648
- [Derived] McNamara B, Demirkiran C, Hartwich TMP, Bellone S, Manavella D, Mutlu L, Greenman M, Zipponi M, Yang-Hartwich Y, Yang K, Ratner E, Schwartz PE, Coma S, Pachter JA, Santin AD. Preclinical efficacy of RAF/MEK clamp avutometinib in combination with FAK inhibition in low grade serous ovarian cancer. Gynecol Oncol. 2024 Apr;183:133-140. doi: 10.1016/j.ygyno.2024.01.028. Epub 2024 Mar 15. PMID 38493021